CLINICAL TRIAL: NCT04961164
Title: A Randomized Double-Blind Cross-over Trial to Study the Effects of Resistant Starch Prebiotic Effects in Chronic Kidney Disease (ReSPECKD)
Brief Title: Resistant Starch Prebiotic Effects in Chronic Kidney Disease
Acronym: ReSPECKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dylan MacKay, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HS23161 (B2019:089)
Record Dates: First submitted 2020-10-26; First posted 2021-07-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease; Resistant Potato Starch; uremic toxins (indoxyl sulphate, p-cresyl sulphate); gut microbiota; metabolomics
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistant Potato Starch (Experimental): 15g RPS mixed with water will be consumed twice per day during intervention
  Interventions: Dietary Supplement: Resistant Potato Starch, Corn Starch
- Corn Starch (Placebo Comparator): 15 g corn starch mixed with water will be consumed twice per day during intervention
  Interventions: Dietary Supplement: Corn Starch, Resistant Potato Starch

INTERVENTIONS:
Dietary Supplement: Resistant Potato Starch, Corn Starch — Consume resistant potato starch at study period 1, then consume corn starch at study period 2.
  Arms: Resistant Potato Starch
Dietary Supplement: Corn Starch, Resistant Potato Starch — Consume corn starch at study period 1, then consume resistant starch at study period 2.
  Arms: Corn Starch

SUMMARY:
In patients with Chronic Kidney Disease (CKD), there is a buildup of nitrogenous uremic toxins of gut microbiome origin, which can contribute to uremic symptoms, reduced quality of life, and earlier progression to dialysis. The goal of this project is to investigate whether the consumption of resistant potato starch (RPS) as an adjunctive therapy to current standard of CKD care will reduce uremic toxins and symptoms by altering the gut microbiota in patients with CKD.

DETAILED DESCRIPTION:
Participants will consent to follow a 18-week study regimen. Participants will receive 2 sachets per day containing either 15 grams of RPS or 15 grams corn starch. The powder in the sachets will be mixed in water and consumed, one sachet in the morning and one before bed. Participants will be instructed to consume the investigational product at least 2 hours prior to or after taking any medication.

For the first two weeks, all participants will go through a run-in period, where they will receive the corn starch. During weeks 3 to 8 (period 1) participants will receive either RPS or cornstarch. The first treatment received will be determined by randomization procedures. During weeks 9 to 12, all participants will undergo a washout period where they will consume cornstarch. During weeks 13 and 18 (period 2), participants will receive the treatment they did not previously consume.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Participant has the ability to speak and read English.
* Male or Female, aged 18 years or above. Females of child-bearing potential must agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include: Hormonal contraceptives including oral contraceptives, hormone birth control patch, vaginal contraceptive ring, injectable contraceptives, or hormone implant, double-barrier method, intrauterine devices, non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s), vasectomy of partner at least 6 months prior to screening.
* Estimated glomerular filtration rate (eGFR) <15 mL/min/1.73m^2 for the past 3 months
* In the Investigator's opinion, participant is able and willing to comply with all trial requirements.

Exclusion Criteria:

* The participant is cognitively impaired and cannot give consent or participate in the group program
* The participant has an existing relationship with the research team, such as supervisory relationship (student, employee) or familial relationship (child, spouse, etc)
* Participants who indicate that they cannot consume study treatments.
* Participants who indicates they are allergic to potatoes or corn
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* History of renal transplant, ongoing dialysis, use of antibiotics (last 3-months), bowel diseases, cancer, surgically removed bowel, or any gastrointestinal surgery (e.g. intestinal resection, gastric bypass, colorectal surgery)
* Inability to consume treatment due to swallowing or GI issues and inability to obtain written informed consent.
* Participating in another interventional trial that could influence the intervention or outcome of this trial.
* Participants with uncontrolled diabetes with a hemoglobin A1C > 10%.
* Participants who consume probiotic supplements.
* Participants with abnormal constrictions of the gastrointestinal tract, diseases of the oesophagus and/or the superior opening of the stomach (cardia), potential or existing intestinal blockage, paralysis of the intestine, megacolon, faecal impaction, appendicitis, a sudden change in bowel habits that has persisted for more than 2 weeks, undiagnosed rectal bleeding, or failure to defaecate following the use of another laxative prod.
* Participants with severe anemia (hemoglobin less than 70).
* Participants taking medications which inhibit peristaltic movement (e.g. opioids,loperamide).
* Participants taking other fiber supplements or able to maintain high fiber/adequate fiber intake through diet.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in blood uremic toxin, indoxyl sulphate, between treatments | between endpoints of each experimental period (week 8 to week 18)
  Change in indoxyl sulphate concentrations in serum
Change in blood uremic toxin, p-cresyl sulphate, between treatments | between endpoints of each experimental period (week 8 to week 18)
  Change in p-cresyl sulphate concentrations in serum

SECONDARY OUTCOMES:
Change in symptoms score using the Edmonton Symptom Assessment Scale between treatments | between endpoints of each experimental period (week 8 to week 18)
  Edmonton Symptom Assessment Scale (ESAS). Minimum value 0 and maximum value 100 with higher values being worse. This assessment will be completed through paper or online by RedCAP.
Change in quality of life of participants between treatments | between endpoints of each experimental period (week 8 to week 18)
  Medical Outcomes Study Short Form 36-item questionnaire (SF-36). This questionnaire will be used as self-reported health and wellness assessment. The scoring ranges from 0 to 100. Higher scores indicate better health status.
Change in alpha diversity of the gut microbiome between treatments | between endpoints of each experimental period (week 8 to week 18)
  Shannon index will be computed to measure of richness and evenness of the Operational Taxonomic Units in each sample
Change in beta diversity of the gut microbiome between treatments | between endpoints of each experimental period (week 8 to week 18)
  Bray-Curtis dissimilarity will be computed to measure microbiome composition similarity among samples
Change in differential abundance in the gut microbiome between treatments | between endpoints of each experimental period (week 8 to week 18)
  Identified Operational Taxonomic Units will be tested for differential abundance using DESeq2 package

OTHER OUTCOMES:
Change in waist circumference | between endpoints of each experimental period (week 8 to week 18)
  Waist circumference will be measured in cm.
Change in body weight | between endpoints of each experimental period (week 8 to week 18)
  Body weight will be measured in kg
Change in serum glucose | between endpoints of each experimental period (week 8 to week 18)
  glucose in mmol/L
Change in Hemoglobin A1c | between endpoints of each experimental period (week 8 to week 18)
  Hemoglobin A1c as percentage
Change in urinary total protein | between endpoints of each experimental period (week 8 to week 18)
  Total protein in mg/dL
Change in urinary glucose concentration | between endpoints of each experimental period (week 8 to week 18)
  Glucose in mmol/L
Change in urinary albumin/creatinine ratio | between endpoints of each experimental period (week 8 to week 18)
  albumin concentration in milligrams divided by creatinine concentration in grams

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Mackay, PhD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Chronic Disease Innovation Centre, Seven Oaks Hospital, Winnipeg, Manitoba
  - Health Science Centre (HSC), Winnipeg, Manitoba

REFERENCES:
- [Derived] Shamloo M, Mollard R, Wang H, Kingra K, Tangri N, MacKay D. A randomized double-blind cross-over trial to study the effects of resistant starch prebiotic in chronic kidney disease (ReSPECKD). Trials. 2022 Jan 24;23(1):72. doi: 10.1186/s13063-022-06009-1. PMID 35073986